CLINICAL TRIAL: NCT05700305
Title: A Feasibility Study to Explore the Role of Exercise and Nutrition to Target Frailty in People With Problematic Substance Use and Homelessness
Brief Title: Physical Rehabilitation Intervention With Protein Supplementation for People With Problematic Substance Use and Homelessness
Status: Completed | Type: Observational
Sponsor: University of Dublin, Trinity College (Other)
Responsible Party: Principal Investigator, Julie Broderick, Assistant Professor, University of Dublin, Trinity College
Other Study IDs: Trinity College Dublin
Record Dates: First submitted 2022-07-19; First posted 2023-01-26 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Social Isolation; Chronic Disease; Physical Disability; Addiction
MeSH Terms: conditions — Social Isolation; Chronic Disease; Behavior, Addictive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: 12-week, low threshold physical rehabilitation intervention with protein supplementation — 12 week, low threshold, rolling exercise intervention with protein supplementation
  Other Names: Physical rehabilitation intervention with protein supplementation

SUMMARY:
Background: People who are homeless are more likely to experience poor mental health and addiction as well as suffering from non-communicable diseases. There is evidence of frailty and accelerated physical ageing among people experiencing homelessness. Appropriate physical rehabilitation and nutritional supplementation strategies can stabilize or reverse frailty and general physical decline, but it is not known how this type of intervention would work in practice in this population.

Aim: To evaluate the feasibility and preliminary efficacy of a physical rehabilitation drop in intervention with protein supplementation to target physical functioning and frailty in people with problematic substance use who are experiencing homelessness.

Methods: The intervention will consist of a 12-week low threshold physical rehabilitation program with protein supplementation. Participants will be service users of the Advance Ballyfermot Project, a day services center for people who are homeless and have active addiction issues. Primary outcomes will be feasibility including numbers recruited, retention of participants and number of repeat visits. Any adverse events will be recorded. Secondary outcomes will be strength and muscular mass, physical performance and lower extremity physical function, pain, frailty and nutritional status.

DETAILED DESCRIPTION:
This single arm feasibility cohort study is taking place in the Advance Ballyfermot Project, located in Dublin. This centre provides a 5-day a week meal service as well as drug related services for people with active addiction issues who are temporarily housed or homeless. A dedicated exercise room has been allocated for the duration of the intervention period. This study has received ethical approval from the Faculty of Health Sciences REC at Trinity College Dublin (Ethical Approval Reference Number: 211202).

The aim of the study is to be as low threshold as possible. This means that minimal constraints are put in place to access the intervention. In order to be as pragmatic as possible in terms of inclusion criteria, all clients (>18 years) accessing services from The Advance Ballyfermot Project who consent to study participation can be included in this study. Only participants with acute problematic behavioral issues or confusion, are in an agitated state or have major physical problems ,(medical or orthopedic) which would preclude ability to safely participate in the exercise class will be excluded from study participation. Participants with a confirmed pregnancy will also be excluded.

The intervention will consist of a twice weekly (for 12 weeks, from November 2022 to February 2023) exercise class with nutritional intervention and a once weekly 'Park Walk'. The intervention will be fully supervised and delivered by two research physiotherapists.

Each session will commence with a warm-up and stretch of the major muscles and will end with cool-down and stretch. The intensity of the workout will be managed by using the Borg Perceived Rate of Exertion (RPE) scale where participants will be advised to exercise at a rate of between 11 and 13 on the PRE scale, ie. between 'fairly light' to 'somewhat hard', where they find it hard to have a conversation but can comfortably continue to exercise.

In an attempt to build sustainability beyond the life cycle of the project, participants will also be educated about exercise and available local resources where possible. Clients will be invited and encouraged to return weekly to continue with the exercise intervention.

The service provided will be low threshold to facilitate adherence and compliance. The research physiotherapists will make every effort to be flexible and accommodating to participants who do not need to make repeat appointments and may turn up on the day of the intervention. Adherence to the program will be measured by the uptake, compliance and number of repeat visits to the drop-in program. Demographic information will include biological sex and current homeless status.

Demographic details, including age, and named General Practitioner (GP) of participants will be collected. A letter will be sent to the GP to inform them of study participation. Questions around current addiction status will be guided by Section 1 of the Treatment Outcome Profile (TOP).

Analytic Plan Our study is very much feasibility focused and not hypothesis driven so formal power calculations are not directly applicable. Prospectively, potential participants that meet the study eligibility criteria will be invited to participate. Descriptive statistics will summarize participant demographics and feasibility measures such as attendance rates. Nominal or ordinal variables will be reported as frequencies and percentages. Continuous variables will be summarized as mean and standard deviation if normally distributed and median and inter-quartile range if non-normally distributed. Data will be tested for normality using the Kolmogorov-Smirnov test and will be compared across timepoints using the general linear model procedure (normally distributed data) and the Friedman's test (non-normally distributed data). As participants will be heterogeneous, data will be sub-stratified and participants will be grouped meaningfully. Free text responses from subjective questions will be reported and organized into topic areas.

ELIGIBILITY:
Inclusion criteria:

• Any person (>18 years) accessing services in Ballyfermot Advance

Exclusion criteria:

* Any person with acute problematic behavioural issues, confusion or major physical problems
* Females with confirmed pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clients accessing services in the Advance Ballyfermot Project (Dublin)
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2022-12-05 (Actual); Study Completion 2023-03-10 (Actual)

PRIMARY OUTCOMES:
Recruitment | October to December 2022
  Number recruited to study
Adverse events | Through to study completion, up to 12 weeks
  Any injuries or incidence will be recorded
Adherence | Through to study completion, up to 12 weeks
  Number of repeat visits

SECONDARY OUTCOMES:
Hand-grip dynamometer | Baseline and 12 weeks
  Strength will be measured using a hand-grip dynamometer
Limb circumference measurement | Baseline and 12 weeks
  Measurement of sarcopenia via mid girth circumference measures of calf and upper arm
The Two Minute Walk Test | Baseline and 12 weeks
  Measurement of walking ability and functional capacity
Numerical Rating Scale | Baseline and 12 weeks
  A unidimensional measure of pain intensity from 0-10, with 0 being zero pain and 10 the worst pain imaginable.
Clinical Frailty Scale | Baseline and 12 weeks
  Each point on the scale is correlated with a description of frailty and a visual chart to aid the tester in classifying frailty from 1 (very fit) to 9 (terminally ill). Higher scores indicate higher levels of frailty.
SHARE Frailty instrument | Baseline and 12 weeks
  The SHARE-FI is a valid tool to measure the level of frailty in individuals aged over 50 years. It consists of quick questions related of the following variables; exhaustion, loss of appetite, walking difficulties and low physical activity. Answers are entered into a freely available web calculator to generate a frailty score and a frailty category of non-frail, pre-frail and frail is generated.
Mini-nutritional assessment | Baseline and 12 weeks
  Assesses nutritional status. The maximum score is 14. A score of 12-14 indicates normal nutritional status; a score between 8 and 11 indicates risk of malnutrition and a score of 7 or less indicates malnourishment.
Body mass Index | Baseline and 12 weeks
  Will be estimated using height (stadiometer) and weight (standardised digital scales)
Self-report open ended questions | Baseline and 12 weeks
  Perceptions about health, physical status and exercise
The 10 Metre Walk Test | Baseline and 12 weeks
  Measurement of walking speed
Single Leg Stance Test | Bseline and 12 weeks
  Measurement of balance and postural control
The 30-Second Chair Stand Test | Baseline and 12 weeks
  Measurement of lower limb strength and endurance
Short Form 12 | Baseline and 12 weeks
  A self-report measure of health used across age, disease and treatment groups. It uses eight domains including physical and social activities, pain, mental health, emotional health, vitality and general health perceptions to measure health. The participant completes a 12 question survey which is scored by the researcher. The minimum possible score is 12 and the maximum possible score is 48. Lower scores indicate better health.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Broderick, Principal Investigator — University of Dublin, Trinity College
Locations (1):
- Trinity College Dublin, University of Dublin, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kennedy F, Murray D, Ni Cheallaigh C, Romero-Ortuno R, Broderick J. Evaluation of a Low-threshold Exercise And Protein supplementation intervention for Women (LEAP-W) experiencing homelessness and addiction: Protocol for a single-arm mixed methods feasibility study. PLoS One. 2025 Feb 6;20(2):e0300412. doi: 10.1371/journal.pone.0300412. eCollection 2025. PMID 39913349
- [Derived] Kennedy F, Ni Cheallaigh C, Romero-Ortuno R, Murray D, Broderick J. Acceptability and utility of a broad test battery to evaluate physical functioning and frailty in community-based settings for people experiencing homelessness and addiction-Findings from the LEAP trials. Physiotherapy. 2025 Mar;126:101449. doi: 10.1016/j.physio.2024.101449. Epub 2024 Nov 7. PMID 39626407